CLINICAL TRIAL: NCT02559505
Title: Understanding How the Initial Encounter With Influenza Virus Poises Children for Protective Immunity
Brief Title: Influenza Immunity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jennifer Nayak, Associate Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RSRB00058437
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Influenza
Keywords: natural influenza infection; live attenuated influenza vaccination (LAIV); inactivated influenza vaccination (IIV); infants; children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 6-12 months Seasonal IIV (Experimental): Children 6 - 12 months of age vaccinated with seasonal IIV
  Interventions: Biological: Seasonal IIV 0.25 mL dose
- 3-12 months natural infection (Experimental): Children 3-12 months of age presenting with natural influenza infection
  Interventions: Other: Natural influenza infection; Biological: Seasonal IIV 0.5 mL dose
- 13-35 months Seasonal IIV (Experimental): Children 13-35 months of age vaccinated with seasonal IIV
  Interventions: Biological: Seasonal IIV 0.25 mL dose
- 13-35 months natural infection (Experimental): Children 13-35 months of age presenting with natural influenza infection
  Interventions: Other: Natural influenza infection; Biological: Seasonal IIV 0.5 mL dose
- 3-5 years Seasonal IIV (Experimental): Children 3-5 years of age vaccinated with seasonal IIV
  Interventions: Biological: Seasonal IIV 0.5 mL dose
- 3-5 years natural infection (Experimental): Children 3-5 years of age presenting with natural influenza infection
  Interventions: Other: Natural influenza infection; Biological: Seasonal IIV 0.5 mL dose
- 6-8 years Seasonal IIV (Experimental): Children 6-8 years of age vaccinated with seasonal IIV
  Interventions: Biological: Seasonal IIV 0.5 mL dose
- 6-8 years natural infection (Experimental): Children 6-8 years of age presenting with natural influenza infection
  Interventions: Other: Natural influenza infection; Biological: Seasonal IIV 0.5 mL dose

INTERVENTIONS:
Biological: Seasonal IIV 0.25 mL dose — Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
  Other Names: Inactivated influenza vaccine
  Arms: 13-35 months Seasonal IIV; 6-12 months Seasonal IIV
Other: Natural influenza infection — Children enrolled on presentation to their primary care provider with a natural influenza infection
  Arms: 13-35 months natural infection; 3-12 months natural infection; 3-5 years natural infection; 6-8 years natural infection
Biological: Seasonal IIV 0.5 mL dose — Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
  Other Names: inactivated influenza vaccine
  Arms: 13-35 months natural infection; 3-12 months natural infection; 3-5 years Seasonal IIV; 3-5 years natural infection; 6-8 years Seasonal IIV; 6-8 years natural infection

SUMMARY:
This study evaluates how different methods of early exposure to influenza (natural infection, live attenuated influenza vaccination, inactivated influenza vaccination) initially stimulate immunity and poise the immune system to respond to a future challenge with the inactivated influenza vaccine.

DETAILED DESCRIPTION:
The proposed research addresses the fact that, despite high childhood morbidity from influenza and broad recommendations for vaccination, very little is known about how anti-influenza immunity is shaped by the method of initial exposure. The objective of this research is to understand how CD4 T cell and B cell responses are altered by the method of initial influenza priming, with the long-term goal of determining how a child's initial influenza encounter poises the immune system to respond to subsequent influenza challenges. The investigators central hypothesis is that differences in the mode of influenza antigen exposure in early childhood will generate long lasting, detectable changes in memory CD4 T cell and B cell specificity and function that influence the response to future influenza vaccinations and infections. This hypothesis will be tested by comparing 1) CD4 T cell and 2) antibody responses in cohorts of children initially exposed to influenza through either natural infection or inactivated or live attenuated vaccination. A combination of multiparameter assays will be used to determine the phenotype and functional potential of hemagglutinin (HA)- and nucleoprotein (NP)-specific CD4 T cells. The breadth and avidity of the neutralizing and non-neutralizing antibody responses and its distribution against head and stalk epitopes will also be evaluated. By determining how initial priming shapes the specificity and functional potential of the anti-influenza CD4 T cell and antibody responses, the investigators will gain the knowledge necessary to optimize current influenza vaccination strategies and develop novel influenza vaccines able to provide highly efficacious universal protection against both seasonal and potentially pandemic viral strains.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * Between 6 and 12 months to participate in the vaccination arm of cohort 1 (cohort 1A)
  * Between 3 and 12 months to participate in the natural infection arm of cohort 1 (cohort 1B)
  * Between 13 and 35 months of age to participate in either the vaccination or natural infection arm of cohort 2
  * Between 36 months and 5 years of age to participate in either the vaccination or natural infection arm of cohort 3
  * Between 6 years and 8 years of age to participate in either the vaccination or natural infection arm of cohort 4
* Gestational age of ≥37 weeks at birth
* Parent/guardian can provide informed consent
* Available for the duration of the study
* History of previous IIV administration ONLY for participation in the vaccination arm of cohorts 2, 3, or 4
* Acute illness documented to be due to influenza virus ONLY for participation in the natural infection arms of cohorts 1-4

Exclusion Criteria:

* Immunosuppression as a result of an underlying illness or condition (including HIV or a primary immunodeficiency syndrome)
* Active neoplastic disease
* Use of potentially immunosuppressive medications currently or within the past year (including chemotherapeutic agents) or chronic (>2 weeks) use of oral or inhaled steroid therapy
* A diagnosis of asthma requiring chronic controller medication
* Previous administration of influenza vaccine in the current influenza season ONLY for subjects receiving an influenza vaccination
* Receipt of immunoglobulin or another blood product within the year prior to study enrollment
* An acute illness within the previous 3 days or temperature >38o on screening EXCEPT for participation in the natural infection arms of cohorts 1-4
* A contraindication to influenza vaccination EXCEPT infants between 3 and 5 months presenting with natural influenza infection whose only contraindication is their current age

Ages: 3 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Nayak, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Shannon I, White CL, Yang H, Nayak JL. Differences in Influenza-Specific CD4 T-Cell Mediated Immunity Following Acute Infection Versus Inactivated Vaccination in Children. J Infect Dis. 2021 Jun 15;223(12):2164-2173. doi: 10.1093/infdis/jiaa664. PMID 33074330

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute: Children enrolled on presentation to their primary care provider with a natural influenza infection.
- Vaccinated: Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
Period: Overall Study
Arm/Group | Acute | Vaccinated
Started | 49 | 84
Completed | 22 | 62
Not Completed | 27 | 22
Not completed — Lost to Follow-up | 23 | 20
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- 6-12 Months of Age: Vaccinated: Children 6 - 12 months of age vaccinated with seasonal IIV
  Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-12 Months of Age: Acute: Children 3-12 months of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 13-35 Months of Age: Vaccinated: Children 13-35 months of age vaccinated with seasonal IIV
  Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 13-35 Months of Age: Acute: Children 13-35 months of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-5 Years of Age: Vaccinated: Children 3-5 years of age vaccinated with seasonal IIV
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-5 Years of Age: Acute: Children 3-5 years of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 6-8 Years of Age: Vaccinated: Children 6-8 years of age vaccinated with seasonal IIV
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 6-8 Years of Age: Acute: Children 6-8 years of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- Total: Total of all reporting groups
Arm/Group | 6-12 Months of Age: Vaccinated | 3-12 Months of Age: Acute | 13-35 Months of Age: Vaccinated | 13-35 Months of Age: Acute | 3-5 Years of Age: Vaccinated | 3-5 Years of Age: Acute | 6-8 Years of Age: Vaccinated | 6-8 Years of Age: Acute | Total
Number analyzed (Participants) | 13 | 8 | 30 | 19 | 18 | 12 | 23 | 9 | 132
Age, Customized [Number; unit: participants] | 13 | 8 | 30 | 19 | 18 | 12 | 23 | 9 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 14 | 8 | 8 | 6 | 10 | 6 | 64
  Male | 4 | 5 | 16 | 11 | 10 | 6 | 13 | 3 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 4 | 0 | 2 | 0 | 3 | 15
  Not Hispanic or Latino | 10 | 8 | 27 | 15 | 18 | 10 | 23 | 6 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 12 | 11 | 0 | 3 | 1 | 5 | 39
  White | 6 | 4 | 10 | 3 | 14 | 8 | 15 | 2 | 62
  More than one race | 2 | 1 | 7 | 3 | 4 | 0 | 7 | 1 | 25
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 8 | 30 | 19 | 18 | 12 | 23 | 9 | 132

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of IFNg+ CD69+ CD4 T Cells Between Acute (H3N2) Infected and Vaccinated Subjects
Description: % H3- and nucleoprotein (NP)-specific CD4 T cells were measured using intracellular cytokine staining
Time Frame: Visit 2 (day 8-14 post enrollment)
Population: 6 acute participants were infected with influenza strains that were not H3 and therefore were not included in the data analyzed for the primary outcome. Only vaccinated participants that age matched to the acute subjects were analyzed, resulting in 16 acutely infected and 28 vaccinated subjects included in the data analysis.
Measure: Mean (Standard Deviation); unit: percentage of T cells
Groups:
- Acute Infected: Children enrolled on presentation to their primary care provider with a natural influenza infection
Arm/Group | Acute Infected | Vaccinated
Number analyzed (Participants) | 16 | 28
percentage of T cells
  Nucleoprotein | .010 (0.0023) | 0.003 (0.0018)
  H3 protein | 0.009 (0.0019) | 0.002 (0.0015)
Statistical Analysis 1: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.005, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated
Statistical Analysis 2: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.024, ANCOVA — p-value for NP reactivity, difference of Acute Infected vs. Vaccinated

2. Primary Outcome: Mean Percent of IFNg+ CD69+ CD4 T Cells Between Acute (H3N2) Infected and Vaccinated Subjects
Description: % H3- and nucleoprotein (NP)-specific CD4 T cells were measured using intracellular cytokine staining
Time Frame: Visit 3 (day 20-28 post enrollment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Acute Infected | Vaccinated
Number analyzed (Participants) | 16 | 28
Percentage of T cells
  Nucleoprotein | 0.012 (0.0025) | 0.003 (0.0017)
  H3 Protein | 0.006 (0.0021) | 0.004 (0.0014)
Statistical Analysis 1: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.408, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated
Statistical Analysis 2: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.004, ANCOVA — p-value for NP reactivity, difference of Acute Infected vs. Vaccinated

3. Primary Outcome: Mean Percent of IFNg+ CD69+ CD4 T Cells Between Acute (H3N2) Infected and Vaccinated Subjects
Description: % H3- and nucleoprotein (NP)-specific CD4 T cells were measured using intracellular cytokine staining
Time Frame: Visit 4 (day of vaccination year 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Acute Infected | Vaccinated
Number analyzed (Participants) | 16 | 28
Percentage of T cells
  Nucleoprotein | 0.003 (0.0030) | 0.003 (0.0018)
  H3 Protein | 0.007 (0.0022) | 0.003 (0.0015)
Statistical Analysis 1: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.991, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated
Statistical Analysis 2: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.334, ANCOVA — p-value for NP reactivity, difference of Acute Infected vs. Vaccinated

4. Primary Outcome: Mean Percent of IFNg+ CD69+ CD4 T Cells Between Acute (H3N2) Infected and Vaccinated Subjects
Description: % H3 protein- and nucleoprotein (NP)-specific CD4 T cells were measured using intracellular cytokine staining
Time Frame: Visit 5 (day 8-14 post-vaccination year 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Acute Infected | Vaccinated
Number analyzed (Participants) | 16 | 28
Percentage of T cells
  Nucleoprotein | 0.010 (0.0031) | 0.003 (0.0018)
  H3 Protein | 0.008 (0.0026) | 0.004 (0.0015)
Statistical Analysis 1: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.226, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated
Statistical Analysis 2: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.036, ANCOVA — p-value for NP reactivity, difference of Acute Infected vs. Vaccinated

5. Primary Outcome: Mean Percent of IFNg+ CD69+ CD4 T Cells Between Acute (H3N2) Infected and Vaccinated Subjects
Description: % H3 Protein- and nucleoprotein (NP)-specific CD4 T cells were measured using intracellular cytokine staining
Time Frame: Visit 6 (day 20-28 post-vaccination year 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of T cells
Arm/Group | Acute Infected | Vaccinated
Number analyzed (Participants) | 16 | 28
Percentage of T cells
  Nucleoprotein | 0.014 (0.0029) | 0.003 (0.0019)
  H3 Protein | 0.008 (0.0024) | 0.007 (0.0015)
Statistical Analysis 1: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.680, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated
Statistical Analysis 2: Comparison: Acute Infected vs Vaccinated; Test type: Other; p = 0.002, ANCOVA — p-value for H3 reactivity, difference of Acute Infected vs. Vaccinated

6. Secondary Outcome: Mean Change in Percent of IFNg+ CD69+ CD4 T Cells Between Vaccinated Subjects in Different Age Subsets
Description: CD4 T cell quantity and specificity will be measured using intracellular cytokine staining. We report here the mean change in percent of cells reactive to the influenza HA protein and H3 protein.
Time Frame: Baseline to day 24 study year 1
Population: Statistical analysis was completed on all patients who attended all six clinical visits in addition to those who had 3 or more visits that had withdrawn later.
Measure: Mean (Standard Deviation); unit: Mean Percent change
Groups:
- Vaccinated Age Subset (6-12 mo): Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 - 12 months.
- Vaccinated Age Subset (13-35 mo): Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 13 - 35 months.
- Vaccinated Age Subset (3-5 yr): Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 3 - 5 years.
- Vaccinated Age Subset (6-8 yr): Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 - 8 years.
Arm/Group | Vaccinated Age Subset (6-12 mo) | Vaccinated Age Subset (13-35 mo) | Vaccinated Age Subset (3-5 yr) | Vaccinated Age Subset (6-8 yr)
Number analyzed (Participants) | 8 | 12 | 14 | 22
Mean Percent change
  HAB | 0.00112 (0.00290) | 0.00497 (0.00966) | 0.00622 (0.01098) | 0.01713 (0.02657)
  H3 | 0.0006729 (0.0017802) | 0.0002589 (0.005017) | 0.0053456 (0.0101449) | 0.001674 (0.008319)

7. Secondary Outcome: Mean Change in Percent of IFNg+ CD69+ CD4 T Cells Between Vaccinated Subjects in Different Age Subsets
Description: as for outcome 6
Time Frame: Baseline to day 24 study year 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Mean Percent Change
Arm/Group | Vaccinated Age Subset (6-12 mo) | Vaccinated Age Subset (13-35 mo) | Vaccinated Age Subset (3-5 yr) | Vaccinated Age Subset (6-8 yr)
Number analyzed (Participants) | 8 | 12 | 14 | 22
Mean Percent Change
  HAB | 0.00552 (0.01436) | 0.00331 (0.01216) | 0.00003 (0.01096) | 0.005698 (0.01729)
  H3 | 0.00350 (0.00372) | 0.00177 (0.00371) | 0.00188 (0.00650) | -0.0017093 (0.01015)

8. Other Pre Specified Outcome: Change From Baseline to Day 10 and Day 24 in PBMC Gene Expression
Description: Changes in PBMC gene expression patterns due to prior influenza exposure will be assessed using RNA-seq analysis
Time Frame: Days 10 and 24 post vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 18 months
Groups:
- 6-12 Months: Vaccinated: Children 6 - 12 months of age vaccinated with seasonal IIV
  Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-12 Months: Acute: Children 3-12 months of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 13-35 Months: Vaccinated: Children 13-35 months of age vaccinated with seasonal IIV
  Seasonal IIV 0.25 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 13-35 Months: Acute: Children 13-35 months of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-5 Years: Vaccinated: Children 3-5 years of age vaccinated with seasonal IIV
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 3-5 Years: Acute: Children 3-5 years of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 6-8 Years: Vaccinated: Children 6-8 years of age vaccinated with seasonal IIV
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
- 6-8 Years: Acute: Children 6-8 years of age presenting with natural influenza infection
  Natural influenza infection: Children enrolled on presentation to their primary care provider with a natural influenza infection
  Seasonal IIV 0.5 mL dose: Fluzone (Sanofi Pasteur) 0.25 mL administered intramuscularly to children between 6 and 35 months of age
Arm/Group | 6-12 Months: Vaccinated | 3-12 Months: Acute | 13-35 Months: Vaccinated | 13-35 Months: Acute | 3-5 Years: Vaccinated | 3-5 Years: Acute | 6-8 Years: Vaccinated | 6-8 Years: Acute
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8 | 0/30 | 0/19 | 0/18 | 0/12 | 0/23 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/30 | 0/19 | 0/18 | 0/12 | 0/23 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/30 | 0/19 | 0/18 | 0/12 | 0/23 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02559505/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT02559505/ICF_001.pdf